CLINICAL TRIAL: NCT02134093
Title: Effects of Dexmedetomidine on Postoperative Cognitive Dysfunction During One-lung Ventilation in Elder Patients -a Single-center, Randomized ,Double-blinded and Controlled Trial
Brief Title: Effects of Dexmedetomidine on Postoperative Cognitive Dysfunction During One-lung Ventilation in Elder Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, YangLu, physician, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Tangdu sedation
Record Dates: First submitted 2014-04-29; First posted 2014-05-08 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Postoperative Confusion
MeSH Terms: interventions — Rocuronium; Dexmedetomidine; Saline Solution; Propofol; Remifentanil; Vecuronium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Normal saline (Placebo Comparator): Continuous pump infusion of normal saline with identical volume, compared with the low dose and high dose group,until the end of surgery
  Interventions: Drug: Induction of anesthesia,midazolam ,sufentanil,etomidate and rocuronium; Drug: Normal saline; Drug: Maintenance of anesthesia , propofol, remifentanil,vecuronium
- High dose group, dexmedetomidine (Experimental): Continuous pump infusion dexmedetomidine at 1μg/kg for 15 minutes before anesthesia induction ,then continuous pump infusion dexmedetomidine at 0.4μg/kg/h until the end of surgery
  Interventions: Drug: Induction of anesthesia,midazolam ,sufentanil,etomidate and rocuronium; Drug: Dexmedetomidine; Drug: Maintenance of anesthesia , propofol, remifentanil,vecuronium
- Low dose group, dexmedetomidine (Experimental): Continuous pump infusion dexmedetomidine at 0.5μg/kg for 15 minutes before anesthesia induction ,then continuous pump infusion dexmedetomidine at 0.2μg/kg/h until the end of surgery
  Interventions: Drug: Induction of anesthesia,midazolam ,sufentanil,etomidate and rocuronium; Drug: Dexmedetomidine; Drug: Maintenance of anesthesia , propofol, remifentanil,vecuronium

INTERVENTIONS:
Drug: Induction of anesthesia,midazolam ,sufentanil,etomidate and rocuronium — Anesthesia induction:midazolam (0.03~0.05 mg/kg), sufentanil(0. 5~0.8 μg/kg), etomidate ( 0.2~0.6mg/kg) and rocuronium(0.6mg/kg)
Drug: Dexmedetomidine — Continuous pump infusion dexmedetomidine at 0.5μg/kg （low dose group）or 1μg/kg （high dose group）for 15 minutes before anesthesia induction，then followed by a continuous pump infusion at 0.2 μg/kg/h（low dose group）or 0.4μg/kg/h（high dose group） until the end of surgery.
  Arms: High dose group, dexmedetomidine; Low dose group, dexmedetomidine
Drug: Normal saline — Continuous pump infusion normal saline with identical volume of dexmedetomidine.
  Arms: Normal saline
Drug: Maintenance of anesthesia , propofol, remifentanil,vecuronium — Continuous infusion of propofol （3~6 mg/kg/h）, remifentanil （0.05~0.3 μg/kg/min）is required to maintain Entropy within 40~60,Mean Arterial Blood Pressure more than 20% of baseline level , Oxygen Saturation more than 90% , airway pressure less than 40 cm H2O, intermittent injection vecuronium （0.05~0.1mg/kg） as needed to maintain muscle relaxation.

SUMMARY:
This study is to explore the effects of dexmedetomidine on postoperative cognitive dysfunction during one-lung ventilation in elder patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Ongoing one-lung ventilation surgery.
* American Society of Anesthesiologists class I to III.
* Aged between 55 and 75 years old.
* Body Mass Index between 18 and 25 kg/m2.

Exclusion Criteria:

* Systolic blood pressure more than 180 mmHg or lower than 90 mmHg,diastolic blood pressure more than 110 mmHg or lower than 60 mmHg.
* Serious heart,liver,kidney, pulmonary, and endocrine disease or serious infection.
* Suspected or confirmed difficult airway.
* History of abnormal anesthesia.
* Suspected of malignant hyperthermia.
* Use of sedative and antidepressant drug or serious alcoholism
* Mini-mental State Examination less than 17.
* Highest academic degree below grade 6 in primary schools
* Patients inability to exchange with serious visual and hearing impairment or mental disability.
* History of shock.
* Carotid artery stenosis and central nervous system disease such as stroke, epilepsy.
* Allergic to investigational products or with other contraindication.
* Participated in other study within 30 days .

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The change in memory | one day before operation, first day after operation
  The change in memory will be evaluated by Controlled Oral Word Association Test ,Semantic Fluency test
Cognitive function | one day before operation, first day after operation
  Cognitive function will be evaluated by Mini-mentalStateExamination,Digit-Symbol Substitution Test ,Trail Making Test
Postoperative anxiety | one day before operation, first day after operation
  Self-evaluation of Depression Symptoms form,Self-Rating Anxiety Scale,Visual analog scales

SECONDARY OUTCOMES:
Heart rate | At the moment of entering operating room ,the moment of intubation，prior to one lung ventilation,10 minutes,30 minutes afer one lung ventilation,the end of operation and the moment of leaving the operating room
Bleeding volume | At the beginning of operation,at the end of operation,up to 24 hours
Total volume of fluid | At the beginning of operation,at the end of operation,up to 24 hours
Duration of one lung ventilation | At the beginning of one lung ventilation,at the end of one lung ventilation,an expected average of 3 hours
The total dose of anaesthetic drugs | At the beginning of surgery,at the end of surgery,up to 24 hours
The total dose of analgesic drugs | During perioperative period,up to 7 days
Blood pressure | At the moment of entering operating room ,the moment of intubation，prior to one lung ventilation,10 minutes,30 minutes afer one lung ventilation,the end of operation and the moment of leaving the operating room
Oxygen saturation | At the moment of entering operating room ,the moment of intubation，prior to one lung ventilation,10 minutes,30 minutes afer one lung ventilation,the end of operation and the moment of leaving the operating room
End-tidal carbon dioxide | At the moment of entering operating room ,the moment of intubation，prior to one lung ventilation,10 minutes,30 minutes afer one lung ventilation,the end of operation and the moment of leaving the operating room
Operation duration | At the beginning of surgery,at the end of surgery,up to 24 hours